CLINICAL TRIAL: NCT00766363
Title: A Randomized, Double-Blind, Placebo-Controlled, Ascending-Dose Phase 1b Safety Study of Three Different Doses of an Alpha-7 Nicotinic Acetylcholine Receptor Agonist (EVP-6124) or Placebo in Patients With Mild to Moderate Probable Alzheimer's Disease
Brief Title: Safety, Tolerability, and Pharmacokinetic Study of EVP-6124 in Patients With Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: FORUM Pharmaceuticals Inc (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EVP-6124-007
Record Dates: First submitted 2008-10-01; First posted 2008-10-03 (Estimated); Results first posted 2011-07-14 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Alzheimer's Disease; Central Nervous System Diseases
Keywords: Alzheimer's Disease; Central Nervous System Diseases; Pharmacokinetics; Cognition
MeSH Terms: conditions — Alzheimer Disease; Central Nervous System Diseases | interventions — 7-chloro-N-quinuclidin-3-yl-benzo(b)thiophene-2-carboxamide; Donepezil; Rivastigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- EVP-6124 (0.1 mg/day) (Experimental)
  Interventions: Drug: EVP-6124 (0.1 mg/day); Drug: Donepezil; Drug: Rivastigmine
- EVP-6124 (0.3 mg/day) (Experimental)
  Interventions: Drug: EVP-6124 (0.3 mg/day); Drug: Donepezil; Drug: Rivastigmine
- EVP-6124 (1.0 mg/day) (Experimental)
  Interventions: Drug: EVP-6124 (1.0 mg/day); Drug: Donepezil; Drug: Rivastigmine
- Placebo (Placebo Comparator)
  Interventions: Drug: Comparator: Placebo; Drug: Donepezil; Drug: Rivastigmine

INTERVENTIONS:
Drug: EVP-6124 (0.1 mg/day) — EVP-6124 was administered as one 0.1 mg capsule per day for 28 days.
  Arms: EVP-6124 (0.1 mg/day)
Drug: EVP-6124 (0.3 mg/day) — EVP-6124 was administered as one 0.3 mg capsule every day for 28 days.
  Arms: EVP-6124 (0.3 mg/day)
Drug: EVP-6124 (1.0 mg/day) — EVP-6124 was administered as one 1.0 mg capsule every day for 28 days.
  Arms: EVP-6124 (1.0 mg/day)
Drug: Comparator: Placebo — Matching placebo was administered as one capsule per day for 28 days.
  Arms: Placebo
Drug: Donepezil — Concomitant therapy with donepezil at a stable dose, taken daily at the same time or immediately after the assigned EVP-6124 dose. Patients must have been taking concomitant therapy for at least 3 months prior to enrollment to be eligible for the study.
Drug: Rivastigmine — Concomitant therapy with rivastigmine at a stable dose, taken daily at the same time or immediately after the assigned EVP-6124 dose. Patients must have been taking concomitant therapy for at least 3 months prior to enrollment to be eligible for the study.

SUMMARY:
This study is being conducted to determine the safety, tolerability, and pharmacokinetics (PK) of three different doses of an investigational medication, EVP-6124, in individuals with mild to moderate Alzheimer's disease who are also taking an Alzheimer's medication (AChEI [acetylcholinesterase inhibitor]: either donepezil or rivastigmine). In addition, PK of AChEI medications will be assessed. Cognitive function will be evaluated on an exploratory basis.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, Phase 1b safety study of three dose levels of EVP-6124 in subjects with mild or moderate Alzheimer's disease and who are taking an AChEI medication (donepezil or rivastigmine).

Study drug will be supplied as capsules and will be orally administered once daily for a total of 28 days. Eligible subjects will be admitted to an inpatient study unit on Day -2 (two days before the first dose of study drug is administered) and will remain confined to the inpatient study unit for a total of five days. Starting on Day 4, subjects will continue the study in the outpatient setting, with study visits on Days 7, 14, 21, and 28. Safety assessments, PK sampling, and cognitive testing will be performed inpatient and at each study visit.

ELIGIBILITY:
Inclusion Criteria:

* male and post-menopausal or surgically sterile female pts
* 50-90 yrs old, who meet clinical criteria for probable Alzheimer's disease (Mini-Mental State Examination of 18-26; Hachinski Ischemic Score ≤4)
* must be taking donepezil or rivastigmine for at least 3 mos.

Exclusion Criteria:

* Unstable medical condition that is clinically significant in the judgment of the investigator; major organ system dysfunction
* Untreated hypothyroidism
* Insufficiently controlled diabetes mellitus
* Diagnosis of major depression requiring antidepressant medications within the last 5 years
* Stroke within 6 months before screening, or concomitant with onset of dementia
* Certain concomitant medications

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R. Hassmann, D.O., Principal Investigator — Comprehensive Clinical Research; Beth Safirstein, M.D., Principal Investigator — MD Clinical; Stephen Thein, Ph.D., Principal Investigator — Pacific Research Network, Inc.; Jeffrey Apter, M.D., Principal Investigator — Global Medical Institutes
Locations (4):
- United States (4):
  - Pacific Research Network, Inc., San Diego, California
  - MD Clinical, Hallandale, Florida
  - Comprehensive Clinical Research, Berlin, New Jersey
  - Global Medical Institutes, LLC, Princeton, New Jersey

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was from September 2008 to February 2009 at 4 study centers in the US (CA, FL, and 2 in NJ).
Pre-assignment Details: 61 subjects were screened and 49 subjects were enrolled.
Groups:
- EVP-6124 (0.1 mg/Day); EVP-6124 (0.3 mg/Day); EVP-6124 (1.0 mg/Day); Placebo: 1 capsule per day for 28 days.
Period: Overall Study
Arm/Group | EVP-6124 (0.1 mg/Day) | EVP-6124 (0.3 mg/Day) | EVP-6124 (1.0 mg/Day) | Placebo
Started | 12 | 13 | 12 (Number randomized.) | 12 (Number randomized.)
SAFETY POPULATION | 12 | 13 | 11 (Decreased by one subject who took placebo instead due to treatment assignment error.) | 13 (Increased by one subject who took placebo due to treatment assignment error.)
PK POPULATION | 12 | 13 | 10 | 13
Completed | 11 | 12 | 12 | 12
Not Completed | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Adverse Event Prior to Randomization | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | EVP-6124 (0.1 mg/Day) | EVP-6124 (0.3 mg/Day) | EVP-6124 (1.0 mg/Day) | Placebo | Total
Number analyzed (Participants) | 12 | 13 | 11 | 13 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 4 | 4 | 18
  >=65 years | 7 | 8 | 7 | 9 | 31
Age Continuous [Mean (Standard Deviation); unit: years] | 68.6 (8.5) | 68.3 (11.1) | 70.2 (12.3) | 72.0 (10.5) | 69.8 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 6 | 8 | 29
  Male | 4 | 6 | 5 | 5 | 20
Region of Enrollment [Number; unit: participants]
  United States | 12 | 13 | 11 | 13 | 49

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of Multiple Doses of EVP-6124 or Placebo in Subjects With Alzheimer's Disease
Description: All adverse experiences spontaneously reported by subject and/or observed by investigator and repeated clinical evaluation of physical examinations, vital signs, 12-lead ECG (electrocardiogram), ambulatory ECG, and laboratory tests (hematology/blood chemistry/urinalysis)
Time Frame: Pre-treatment (Day -2) [or screening for physical examination] to Day 28 [or Day 35, for AEs only]
Population: Safety Population: All randomized subjects who ingested at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | EVP-6124 (0.1 mg/Day) | EVP-6124 (0.3 mg/Day) | EVP-6124 (1.0 mg/Day) | Placebo
Number analyzed (Participants) | 12 | 13 | 11 | 13
Participants
  Serious Adverse Events | 0 | 0 | 0 | 0
  Non-Serious Adverse Events | 2 | 3 | 4 | 4
  No Adverse Events Reported | 10 | 10 | 7 | 9

2. Secondary Outcome: EVP-6124 PK Data Following the First Dose of EVP-6124 - Maximum Concentration (Cmax)
Description: EVP-6124 PK data; Maximum Concentration (Cmax); i.e, highest concentration of drug in plasma
Time Frame: 24 hours
Population: PK Population: All safety population subjects who had sufficient plasma concentration data to facilitate calculation of PK parameters.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | EVP-6124 (0.1 mg/Day) | EVP-6124 (0.3 mg/Day) | EVP-6124 (1.0 mg/Day)
Number analyzed (Participants) | 12 | 13 | 10
ng/mL | 0.0715 (0.0121) | 0.1911 (0.0740) | 0.6122 (0.1235)

3. Secondary Outcome: EVP-6124 PK Data Following the First Dose of EVP-6124 - Time to Maximum Concentration (Tmax)
Description: EVP-6124 PK data; Time to Maximum Concentration (Tmax); i.e, amount of time required to reach highest concentration of drug in plasma
Time Frame: 24 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | EVP-6124 (0.1 mg/Day) | EVP-6124 (0.3 mg/Day) | EVP-6124 (1.0 mg/Day)
Number analyzed (Participants) | 12 | 13 | 10
hours | 7.70 (3.31) | 7.94 (3.61) | 10.72 (6.69)

4. Secondary Outcome: EVP-6124 PK Data Following the First Dose of EVP-6124 - Area Under the Curve (AUC[0-24 h])
Description: EVP-6124 PK data; Area Under the Curve (AUC[0-24 h]); i.e, area under the concentration-time plot
Time Frame: 24 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | EVP-6124 (0.1 mg/Day) | EVP-6124 (0.3 mg/Day) | EVP-6124 (1.0 mg/Day)
Number analyzed (Participants) | 12 | 11 | 7
h*ng/mL | 1.31 (0.23) | 3.89 (0.84) | 11.44 (2.24)

5. Secondary Outcome: Donepezil PK Data Following the First Dose of EVP-6124 - Maximum Concentration (Cmax)
Description: Donepezil PK data; Maximum Concentration (Cmax); i.e, highest concentration of donepezil (parent compound only) in plasma after dosing with EVP-6124
Time Frame: 24 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | EVP-6124 (0.1 mg/Day) | EVP-6124 (0.3 mg/Day) | EVP-6124 (1.0 mg/Day) | Placebo
Number analyzed (Participants) | 10 | 13 | 7 | 13
ng/mL | 29.5 (15.8) | 24.7 (19.8) | 39.2 (26.7) | 41.9 (19.7)

6. Secondary Outcome: Donepezil PK Data Following the First Dose of EVP-6124 - Time to Maximum Concentration (Tmax)
Description: Donepezil PK data; Time to Maximum Concentration (Tmax); i.e, amount of time required to reach highest concentration of donepezil (parent compound only) in plasma after dosing with EVP-6124
Time Frame: 24 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | EVP-6124 (0.1 mg/Day) | EVP-6124 (0.3 mg/Day) | EVP-6124 (1.0 mg/Day) | Placebo
Number analyzed (Participants) | 10 | 12 | 7 | 13
hours | 2.30 (2.65) | 1.85 (2.15) | 3.31 (3.01) | 3.56 (4.02)

7. Secondary Outcome: Donepezil PK Data Following the First Dose of EVP-6124 - Area Under the Curve (AUC[0-24 h])
Description: Donepezil PK data; Area Under the Curve (AUC[0-24 h]); i.e, area under the concentration-time plot for donepezil (parent compound only) after dosing with EVP-6124
Time Frame: 24 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | EVP-6124 (0.1 mg/Day) | EVP-6124 (0.3 mg/Day) | EVP-6124 (1.0 mg/Day) | Placebo
Number analyzed (Participants) | 10 | 13 | 7 | 13
h*ng/mL | 299 (179) | 240 (194) | 345 (225) | 427 (233)

8. Secondary Outcome: Rivastigmine PK Data Following the First Dose of EVP-6124 - Maximum Concentration (Cmax)
Description: Rivastigmine PK data; Maximum Concentration (Cmax); i.e, highest concentration of rivastigmine in plasma after dosing with EVP-6124
Time Frame: 24 hours
Population: PK Population: All safety population subjects who had sufficient plasma concentration data to facilitate calculation of PK parameters. Only 4 subjects took rivastigmine concomitantly.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | EVP-6124 (0.1 mg/Day) | EVP-6124 (1.0 mg/Day)
Number analyzed (Participants) | 2 | 2
ng/mL | 23.35 (5.16) | 3.51 (0.37)

9. Secondary Outcome: Rivastigmine PK Data Following the First Dose of EVP-6124 - Time to Maximum Concentration (Tmax)
Description: Rivastigmine PK data; Time to Maximum Concentration (Tmax); i.e, amount of time required to reach highest concentration of rivastigmine in plasma after dosing with EVP-6124
Time Frame: 24 hours
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | EVP-6124 (0.1 mg/Day) | EVP-6124 (1.0 mg/Day)
Number analyzed (Participants) | 2 | 2
hours | 1.00 (0.02) | 12.12 (15.72)

10. Secondary Outcome: Rivastigmine PK Data Following the First Dose of EVP-6124 - Area Under the Curve (AUC[0-24 h])
Description: Rivastigmine PK data; Area Under the Curve (AUC[0-24 h]); i.e, area under the concentration-time plot for rivastigmine after dosing with EVP-6124
Time Frame: 24 hours
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | EVP-6124 (0.1 mg/Day) | EVP-6124 (1.0 mg/Day)
Number analyzed (Participants) | 2 | 2
h*ng/mL | 143.55 (85.52) | 54.60 (6.28)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from pre-treatment (Day -2) to 7 days after the last dose of study drug (Day 35).
Arm/Group | EVP-6124 (0.1 mg/Day) | EVP-6124 (0.3 mg/Day) | EVP-6124 (1.0 mg/Day) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13 | 0/11 | 0/13
Other Adverse Events (participants affected / at risk) | 2/12 | 3/13 | 4/11 | 4/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EVP-6124 (0.1 mg/Day) (N=12) | EVP-6124 (0.3 mg/Day) (N=13) | EVP-6124 (1.0 mg/Day) (N=11) | Placebo (N=13)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 60 days from the time submitted for review. At the sponsor's request, the PI will delete confidential information other than trial data and will delay publication or disclosure for up to 90 days to allow patent filings. The PI agrees that the first publication shall be a joint publication.